CLINICAL TRIAL: NCT05357053
Title: Anorexia Nervosa and Its Effects on Brain Function, Body Metabolism and Their Interaction in Adolescents
Acronym: AVAIN_JR
Status: Active, not recruiting | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other)
Responsible Party: Sponsor
Other Study IDs: T163_2021
Record Dates: First submitted 2022-03-28; First posted 2022-05-02 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-04

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia nervosa; Metabolism; Functional Imaging; Eating disorders
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and fecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Anorexia nervosa patients: Anorexia nervosa patients
- Healthy normal weight controls: Healthy normal weight controls

SUMMARY:
The aim of the research project is to investigate the neurological, physiological and behavioral underpinnings associated with the development of anorexia nervosa in adolescents. The goal of the project is to enable new ways to both predict the course of the disease and to influence this process.

DETAILED DESCRIPTION:
The aim of the project is to enable new ways to both predict and influence the course of anorexia nervosa. This is a three-year follow-up study in which we investigate the neurological and physiological factors underpinnings of anorexia nervosa with structural and functional magnetic resonance imaging (fMRI). In addition to this, a variety of methods is used, such as physiological measurements and questionnaire data, as well as investigation of intestinal microbiota associated with anorexia nervosa. Altogether 100 girls aged 13-17 will be recruited for the study: 50 patients with anorexia nervosa and 50 healthy controls. The participants are monitored annually and the fMRI scan is repeated at the last visit. Additionally, 40 participants (20 patients and 20 healthy controls) will participate in a cardiac sub-study. In this, the participants will also have an MRI scan and ultrasound examination of the heart.

ELIGIBILITY:
Inclusion criteria for anorexia nervosa patients:

* Female sex
* Age 13-17 years
* Body mass index < 17.5 kg/m2
* Currently fulfilling modified Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) diagnosis criteria for anorexia nervosa with or without amenorrhea
* Anorexia nervosa diagnosed within 2 yers

Inclusion criteria for healthy controls:

* Female sex
* Age 13-17 years
* Body mass index 18,5-25 kg/m2
* No lifetime history of obesity (Body mass index ≥ 30) or eating disorders

Exclusion criteria:

* Any chronic illness or medication that could affect glucose metabolism or neurotransmission
* Any other current mental disorder (excluding anorexia nervosa for the patient participants)
* Severe previous mental disorder (excluding anorexia nervosa for the patient participants)
* Smoking of tobacco, snuffing, or use of narcotics
* Abusive use of alcohol

Ages: 13 Years to 17 Years | Sex: Female
Age Groups: Child
Study Population: The study population comprises 50 female adolescents with anorexia nervosa meeting the inclusion criteria. They are compared with 50 age and sex-matched healthy normal weight controls.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in brain reward system and metabolism in anorexia nervosa patients | 3 years
  Anorexia nervosa patients and controls are studied using fMRI imaging and followed up for 3 years. Reward system function is measured using fMRI and metabolism using blood oxygen level-dependent (BOLD) echo-planar imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Max Karukivi, MD, PhD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku PET Centre, Turku, Finland